CLINICAL TRIAL: NCT04147923
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Study to Investigate the Effect of Floradapt Mature Immune Defense on Nutrient Uptake and Digestive Health in a Healthy Elderly Population
Brief Title: A Study Investigating the Effect of Floradapt Mature Immune Defense on Nutrient Uptake and Digestive Health in a Healthy Elderly Population
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kaneka Americas Holding Inc. (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 19ANHK
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-01

CONDITIONS: Healthy
Keywords: Probiotic; Digestive Health; Healthy; Nutrient analysis; Constipation
MeSH Terms: conditions — Constipation | interventions — Geritol

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Floradapt Mature Immune Defense (Active Comparator): A multivitamin will also be consumed.
  Interventions: Dietary Supplement: Floradapt Mature Immune Defense + Multivitamin
- Placebo (Placebo Comparator): A multivitamin will also be consumed.
  Interventions: Dietary Supplement: Placebo + Multivitamin

INTERVENTIONS:
Dietary Supplement: Floradapt Mature Immune Defense + Multivitamin — The product consists of two L. plantarum strains, KABP XXXX and KABP XXXX with a combined strength of >1 x 10^9 CFU. Participants will also consume a multivitamin.
  Arms: Floradapt Mature Immune Defense
Dietary Supplement: Placebo + Multivitamin — No active ingredients + a multivitamin supplement
  Arms: Placebo

SUMMARY:
This trial will be investigating the effect for Floradapt Mature Immune Defense on nutrient uptake and digestive health in a healthy elderly population. Approximately 120 healthy older adults will be enrolled into the study and will consume either the probiotic or placebo supplement for 84 days and complete questionnaires as well as provide blood samples for nutrient uptake analysis (for 50 participants), immunological markers, and general markers of health. Saliva samples will be provided for analysis of sIgA and cortisol.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 50 to 85 years, inclusive
2. BMI 18.5-29.9 kg/m2, inclusive
3. Participants must meet the following criteria regarding their bowel habits. This will be assessed at screening and confirmed at baseline:

   I. ≤ 5 complete BMs per week AND at least 25% of BMs are BSS type 1 or 2 collectively with excessive straining for most of the BMs (≥50%), defined as 3 minutes or more during BM, as assessed by the QI OR, II. At least 50% of bowel movements are Bristol Stool Scale (BSS) type 1 and 2 at screening and confirmed at baseline as assessed by the QI OR, III. ≤ 3 complete spontaneous BMs per week as assessed by the QI
4. Female participant is not of child bearing potential, which is defined as females who have had a hysterectomy or bilateral oophorectomy, complete endometrial ablation, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation) OR,

   Females of child-bearing potential must have a negative urine pregnancy test at screening and baseline and must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. A minimum of 3-months stable dose is required for females on a hormonal birth control. Acceptable methods of birth control include:

   I. Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System) II. Double-barrier method III. Intrauterine devices IV. Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s) V. Vasectomy of partner (shown successful as per appropriate follow-up)
5. Albumin levels at screening between 25-50 g/L, inclusive. If albumin level <35 g/L all other liver function tests must be within the normal range.
6. Healthy as determined by laboratory results, medical history, and physical exam by QI
7. Agrees to comply with all study procedures
8. Agrees to maintain current level of physical activity and diet throughout the study

Exclusion Criteria:

1. Women who are pregnant, breast feeding, or planning to become pregnant during the trial
2. Allergy or sensitivity to investigational product's active or inactive ingredients or milk
3. Chronic constipation
4. On prescribed laxatives
5. Current or history of clinically significant diseases of the gastrointestinal tract (examples include but are not limited to atrophic gastritis, celiac disease, gluten intolerance/sensitivity, inflammatory bowel disease)
6. Current or history of pancreatitis or short bowel syndrome
7. Current or history of malabsorption assessed by the QI
8. Major surgery in the past 3 months or individuals who have planned surgery during the course of the trial. Minor surgery will be considered on a case by case basis by QI
9. Cancer, except skin cancers completely excised with no chemotherapy or radiation with a follow up that is negative. Cancer in full remission for more than five years after diagnosis are acceptable.
10. Verbal confirmation of autoimmune disease or if immune-compromised
11. Verbal confirmation of HIV, hepatitis B/C positive diagnosis
12. Current or history of hypertension but on a stable dose medication for ≥ 2 months will be reviewed on a case-by-case basis by the QI.
13. Type I or type II diabetes or use of diabetes medication
14. Significant cardiovascular event in the past 6 months. No significant cardiovascular event on stable medication may be included after assessment by the QI on a case by case basis
15. History or currently with kidney and liver diseases assessed by QI on a case by case basis, with the exception of kidney stone history in participants who are symptom free for 1 year
16. Verbal confirmation of current or pre-existing thyroid condition. Treatment on a stable dose medication for over 3 months will be reviewed on a case-by-case basis by the QI
17. Difficulties swallowing medications
18. Verbal confirmation of bleeding disorder
19. Blood disorders as determined by laboratory results
20. Acute or chronic illness of concern to the QI
21. Clinically significant abnormal laboratory results at screening as assessed by QI
22. Current use of blood thinners, with the exception of ASA 81 mg or less
23. Current use of prescribed medications that may cause constipation or affect the study outcomes as assessed by QI
24. Use of over-the-counter (OTC) medications or supplements or consumption of foods/drinks that may affect the study outcomes, unless willing to undergo an appropriate washout period prior to baseline is agreed upon after assessment by the QI.
25. Medicinal use of marijuana
26. Recreational use of marijuana, unless willing to undergo a 30-day washout prior to baseline
27. Alcohol or drug abuse (< 1 year)
28. High alcohol intake (average of >2 standar3d drinks per day or >10 standard drinks per week)
29. Use of narcotics
30. Illicit drug use in the past 6 months as assessed by the QI
31. Current uses of tobacco or related products unless cessation 60 days prior to baseline
32. Blood donation during or within 30 days following conclusion of clinical trial
33. Participation in a clinical research trial within 30 days prior to enrollment will be assessed case-by-case by the QI
34. Verbal confirmation of dementia or known neuropsychological condition that, in the QI's opinion, could interfere with study participation.
35. Individuals who are cognitively impaired and/or who are unable to give informed consent
36. Any other chronic or active or unstable medical condition, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
The changes from baseline to day 42 between Floradapt Mature Immune Defense and placebo in digestive health as assessed by Gastrointestinal Symptoms Rating Scale (GSRS) | 42 days
  Five symptom clusters depicted as Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation will be assessed from the combination of the 15 items in the questionnaire (Abdominal pains, Heartburn, Acid regurgitation, Sucking sensations in the epigastrium, Nausea and vomiting, Borborygmus, Abdominal distension, Eructation, Increased flatus, Decreased passage of stools, Increased passage of stools, Loose stools, Hard Stools, Urgent need for defecation, Feeling of incomplete evacuation). All the domains will be scored on a 4-point scale where 0 represented no symptoms and 3 represented severe symptoms. A lower score represents less symptoms.
The changes from baseline to day 84 between Floradapt Mature Immune Defense and placebo in digestive health as assessed by Gastrointestinal Symptoms Rating Scale (GSRS) | 84 days
  Five symptom clusters depicted as Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation will be assessed from the combination of the 15 items in the questionnaire (Abdominal pains, Heartburn, Acid regurgitation, Sucking sensations in the epigastrium, Nausea and vomiting, Borborygmus, Abdominal distension, Eructation, Increased flatus, Decreased passage of stools, Increased passage of stools, Loose stools, Hard Stools, Urgent need for defecation, Feeling of incomplete evacuation). All the domains will be scored on a 4-point scale where 0 represented no symptoms and 3 represented severe symptoms. A lower score represents less symptoms.
The changes from baseline to day 42 between Floradapt Mature Immune Defense and placebo in bowel movements and stool consistency as assessed by daily bowel habits diary | 42 days
  The Bowel Habit Diary consisted of a 7 items questionnaire for evaluating each bowel movement. Bristol Stool Scale is a seven-stool description and image scale within the Daily Bowel Habit Diary to assess stool shape and consistency (type 1 is separate hard lumps, where type 7 is watery stools with no solid pieces). Stool consistency is a bowel function indicator due to its correlation with colonic transit time.
The changes from baseline to day 84 between Floradapt Mature Immune Defense and placebo in bowel movements and stool consistency as assessed by daily bowel habits diary | 84 days
  The Bowel Habit Diary consisted of a 7 items questionnaire for evaluating each bowel movement. Bristol Stool Scale is a seven-stool description and image scale within the Daily Bowel Habit Diary to assess stool shape and consistency (type 1 is separate hard lumps, where type 7 is watery stools with no solid pieces). Stool consistency is a bowel function indicator due to its correlation with colonic transit time.
The changes from baseline to day 42 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing serum levels of albumin | 42 days
The changes from baseline to day 84 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing serum levels of albumin | 84 days
The changes from baseline to day 42 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing serum levels of total protein | 42 days
The changes from baseline to day 84 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing serum levels of total protein | 84 days
The changes from baseline to day 42 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing serum levels of Vitamin A | 42 days
The changes from baseline to day 84 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing serum levels of Vitamin A | 84 days
The changes from baseline to day 42 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing serum levels of Vitamin B12 | 42 days
The changes from baseline to day 84 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing serum levels of Vitamin B12 | 84 days
The changes from baseline to day 42 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing serum levels of Folate | 42 days
The changes from baseline to day 84 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing serum levels of Folate | 84 days
The changes from baseline to day 42 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing serum levels of Vitamin C | 42 days
The changes from baseline to day 84 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing serum levels of Vitamin C | 84 days
The changes from baseline to day 42 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing serum levels of Vitamin D | 42 days
The changes from baseline to day 84 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing serum levels of Vitamin D | 84 days
The changes from baseline to day 42 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing serum levels of Vitamin E | 42 days
The changes from baseline to day 84 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing serum levels of Vitamin E | 84 days
The changes from baseline to day 42 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing serum levels of Calcium | 42 days
The changes from baseline to day 84 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing serum levels of Calcium | 84 days
The changes from baseline to day 42 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing serum levels of Iron | 42 days
The changes from baseline to day 84 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing serum levels of Iron | 84 days
The changes from baseline to day 42 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing serum levels of Magnesium | 42 days
The changes from baseline to day 84 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing serum levels of Magnesium | 84 days
The changes from baseline to day 42 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing plasma levels of Vitamin B6 | 42 days
The changes from baseline to day 84 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing plasma levels of Vitamin B6 | 84 days
The changes from baseline to day 42 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing plasma levels of Zinc | 42 days
The changes from baseline to day 84 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing plasma levels of Zinc | 84 days
The changes from baseline to day 42 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing plasma levels of CoQ10 | 42 days
The changes from baseline to day 84 between Floradapt Mature Immune Defense and placebo in nutrient uptake as determined by analyzing plasma levels of CoQ10 | 84 days

SECONDARY OUTCOMES:
The change from baseline to day 84 between Floradapt Mature Immune Defense and placebo in quality of life (QoL) assessed by the SF-12v2 questionnaire | 84 days
The change from baseline to day 84 between Floradapt Mature Immune Defense and placebo in quality of life (QoL) assessed by Perceived Stress test | 84 days
The changes in plasma immunological marker CD4+from baseline to day 42 between Floradapt Mature Immune Defense and placebo supplementation | 42 days
The changes in plasma immunological marker CD4+from baseline to day 84 between Floradapt Mature Immune Defense and placebo supplementation | 84 days
The changes in plasma immunological marker CD8+from baseline to day 42 between Floradapt Mature Immune Defense and placebo supplementation | 42 days
The changes in plasma immunological marker CD8+from baseline to day 84 between Floradapt Mature Immune Defense and placebo supplementation | 84 days
The changes in plasma immunological marker CD19+ from baseline to day 42 between Floradapt Mature Immune Defense and placebo supplementation | 42 days
The changes in plasma immunological marker CD19+ from baseline to day 84 between Floradapt Mature Immune Defense and placebo supplementation | 84 days
The changes in plasma immunological marker CD56+ from baseline to day 42 between Floradapt Mature Immune Defense and placebo supplementation | 42 days
The changes in plasma immunological marker CD56+ from baseline to day 84 between Floradapt Mature Immune Defense and placebo supplementation | 84 days
The changes in saliva immunological marker sIgA from baseline to day 42 between Floradapt Mature Immune Defense and placebo supplementation | 42 days
The changes in saliva immunological marker sIgA from baseline to day 84 between Floradapt Mature Immune Defense and placebo supplementation | 84 days
The changes in saliva immunological marker cortisol from baseline to day 42 between Floradapt Mature Immune Defense and placebo supplementation | 42 days
The changes in saliva immunological marker cortisol from baseline to day 84 between Floradapt Mature Immune Defense and placebo supplementation | 84 days

OTHER OUTCOMES:
Incidence of pre-emergent and post-emergent adverse events following 84-day between Floradapt Mature Immune Defense and placebo supplementation | 84 days
The change in systolic blood pressure when supplemented for 84-days with either Floradapt Mature Immune Defense or placebo | 84 days
The change in diastolic blood pressure when supplemented for 84-days with either Floradapt Mature Immune Defense or placebo | 84 days
The change in heart rate when supplemented for 84-days with either Floradapt Mature Immune Defense or placebo | 84 days
The change in alanine aminotransferase (ALT) following 84-day supplementation with Floradapt Mature Immune Defense or placebo | 84 days
The change in aspartate aminotransferase (AST) following 84-day supplementation with Floradapt Mature Immune Defense or placebo | 84 days
The change in total bilirubin following 84-day supplementation with Floradapt Mature Immune Defense or placebo | 84 days
The change in creatinine following 84-day supplementation with Floradapt Mature Immune Defense or placebo | 84 days
The change in electrolytes following 84-day supplementation with Floradapt Mature Immune Defense or placebo | 84 days
The change in estimated glomerular filtration rate (eGFR) following 84-day supplementation with Floradapt Mature Immune Defense or placebo | 84 days
The change in neutrophils after 84-day supplementation with Floradapt Mature Immune Defense or placebo | 84 days
The change in lymphocytes after 84-day supplementation with Floradapt Mature Immune Defense or placebo | 84 days
The change in monocytes after 84-day supplementation with Floradapt Mature Immune Defense or placebo | 84 days
The change in eosinophils after 84-day supplementation with Floradapt Mature Immune Defense or placebo | 84 days
The change in basophils after 84-day supplementation with Floradapt Mature Immune Defense or placebo | 84 days
The change in red blood cell (RBC) count after 84-day supplementation with Floradapt Mature Immune Defense or placebo | 84 days
The change in hemoglobin levels after 84-day supplementation with Floradapt Mature Immune Defense or placebo | 84 days
The change in hematocrit levels after 84-day supplementation with Floradapt Mature Immune Defense or placebo | 84 days
The change in platelet count after 84-day supplementation with Floradapt Mature Immune Defense or placebo | 84 days
The change in mean corpuscular volume (MCV) after 84-day supplementation with Floradapt Mature Immune Defense or placebo | 84 days
The change in mean corpuscular hemoglobin (MCH) after 84-day supplementation with Floradapt Mature Immune Defense or placebo | 84 days
The change in mean corpuscular hemoglobin concentration (MCHC) after 84-day supplementation with Floradapt Mature Immune Defense or placebo | 84 days
The change in mean platelet volume (MPV) after 84-day supplementation with Floradapt Mature Immune Defense or placebo | 84 days
The change in red cell distribution width (RDW) after 84-day supplementation with Floradapt Mature Immune Defense or placebo | 84 days

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh RG, Aoki F, Rodriguez-Palmero Seuma M, Aguilo M, Washida M, Espadaler-Mazo J, Al-Wahsh H, Crowley DC, Guthrie N, Evans M, Moulin M, Lewis ED. Efficacy of Probiotic Supplementation with Lactiplantibacillus plantarum Strains on Gastrointestinal Tract Function - A Randomized Controlled Trial. J Diet Suppl. 2025;22(4):549-570. doi: 10.1080/19390211.2025.2507610. Epub 2025 Jun 4. PMID 40468693